CLINICAL TRIAL: NCT05891704
Title: The Efficacy of Hand Injuries Rehabilitation Intervention Program That Incorporated Ethnic and Cultural Reference
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Navah Ratzon, Head of School of Health Profession, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Jumana Daibes
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Injuries of Hand (Disorder)
Keywords: Hand Injury, Values, Culture, ACT, Hand Injury Intervention
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Intervention Group (IG) will receive 12-16 meetings of the standard conventional hand-therapy program according to OT intervention protocols used for clients with HI. The IG will receive one hour of 2-3 sessions a week according to patient needs and convenience. In each treatment session, the participant will receive 30 minutes of preparatory activities and therapeutic exercise, 15 min of Occupation-Based Activities, and 15 min for the culturally adjusted intervention that will be based on Focused Acceptance and Commitment Therapy (FACT) with major emphasis on values. In IG Arabic cultural values will be considered in the entire therapy process, the participant will have a companion in the therapy session. The participants in IG will be provided with a home-therapy protocol, and will complete a home program that will be based on enhancement of work values. Checklist diary will be provided to participants
  Interventions: Procedure: Hand therapy Rehabilitation intervention program that incorporate cultural reference
- Control group (Active Comparator): The Control Group (CG) will follow the identical therapy protocol as the IG which will last for 45 minutes, with no culturally relevant interventions. In addition, each participant in the CG group will receive 15 minutes of free conversation with narrative feedback regarding the therapy, the challenges and opportunities in his daily life. Home-therapy protocol that will be based on conventional intervention will be provided.
  Interventions: Procedure: Conventional Hand therapy Rehabilitation intervention program

INTERVENTIONS:
Procedure: Hand therapy Rehabilitation intervention program that incorporate cultural reference — The intervention will provide a conventional hand therapy rehabilitation intervention program that incorporates cultural reference based on Focused Acceptance and commitment Therapy ( FACT).
  Arms: Intervention group
Procedure: Conventional Hand therapy Rehabilitation intervention program — The intervention will provide a conventional hand therapy rehabilitation intervention program
  Arms: Control group

SUMMARY:
The study has three main phases. The first phase included A. Adjustment of research tools. Phase B. will examine the efficacy of the cultural intervention. Phase C. Follow-up study will be conducted after three, six, and nine months.

DETAILED DESCRIPTION:
Trauma to the hand is a common and potentially serious injury. Work is central to most adults' occupational identity and is, therefore, a key focus for occupational therapy (OT) intervention. There is substantial evidence that supports the use of OT to target work and its positive influence on Return to Work (RTW) after injury. OT literature shows a shift regarding the awareness of cultural concerns and the broader context in which OT operates. There is currently no high-quality evidence to support the efficacy of rehabilitation programs that enhance RTW in workers with Hand Injury (HI). Aims: The proposed study aims to examine the efficacy of a hand-injuries rehabilitation intervention program that incorporates ethnic-cultural references versus conventional intervention programs. Objective and subjective measures will be used to evaluate personal and environmental aspects and address their influence on readiness to RTW, time to RTW, and, for those who will RTW, employer satisfaction about the worker's performance. Method: The Study has Three Phases: 1. A cross-sectional study to assess internal consistency and test-retest reliability and construct and concurrent validity of the study questionnaires. Study participants: Convenient sample of 60 healthy and 30 HI Palestinian participants will be recruited. Tools: Arabic Work Value Questionnaire (A-Wval), the Arabic Employment Barrier Questionnaire (A-EBQ), the Arabic Return to Work Self-Efficacy-19 (A-RTWSE-19) questionnaire, the Arabic Readiness for Return-To-Work (A-RRTW), Arabic Return-to-Work status questionnaire (A-RTWS), and Arabic Work Behavior Inventory (A-WBI). 2. Matched paired trial design method will be conducted to assess the efficacy of a hand-injuries rehabilitation intervention program that incorporates ethnic-cultural reference versus conventional intervention programs that will improve the participants' functioning in Vocational Rehabilitation(VR) and enhance Time of Return to Work (TRTW). Study participants: 100 HI participants will be first matched in pairs according to gender, age (interval of 5 years), and severity of the injury. Then, each member of a pair will be randomly assigned to the intervention group (IG) and Control Group (CG). 3. Follow-up study after three, six, and nine months.

ELIGIBILITY:
Inclusion Criteria: Participants will include people after acute traumatic injuries below the elbow, 16-65 years old, who were employed or functioning as active housewives prior to the injury. All participants will be Palestinian Arabs living in the West Bank

Exclusion Criteria: People with drug/alcohol abuse, central nervous lesions, psychiatric, cognitive or developmental disorder, people with bilateral injury, hand burns, rheumatoid arthritis, osteoarthritis, brachial plexus lesion, shoulder or elbow problems, complex regional pain syndrome, or any surgery during the study period. People with non-traumatic hand injuries (tendonitis, carpal tunnel syndrome, trigger finger, De Quervain's disease, and Mallet finger) will not be included

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
A change in baseline of Time to Return to Work (T-RTW) to discharge from therapy and the change at three, six, and nine months are being assessed. | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  the time to return to work since onset
A change in a baseline evaluation of the Disabilities of the Arm, Shoulder, and Hand questionnaire (Quick DASH) to discharge and from therapy and the change at three, six, and nine months are being assessed. | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  The self-reported upper extremity outcome measure for assessing physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb, whose primary language is Arabic.
A change in baseline Work Rehabilitation Questionnaire (WORQ) (Finger, Escorpizo, Bostan, & De Bie, 2014) to discharge from therapy and at three, six, and nine months follow-up is being assessed. | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  ICF-based questionnaire to evaluate functioning in Vocational Rehabilitation (VR), The WORQ consists of two sections. Section 1 contains 17 socio demographic and work-related items, the work-related questions include profession, work status, work demands, VR interventions, and the amount of support received by family, employer, and labor and employment services while section two contains 40 items on functioning (18 body functions and 22 activities and participation items). WORQ captures the extent of functioning problems for all 40 items with a numeric rating scale of 0 to 10

SECONDARY OUTCOMES:
Modified Hand Injury Scoring System (MHISS) (Campbell & Kay, 1996; Urso-Baiarda et al., 2008) | Baseline Time (T1)
  MHISS is an objective anatomical assessment specifically designed for hand injuries. The hand injuries can be divided into four broad categories, such as "Minor" (< 20 moderate (21-50 points), severe (51-100 points), and major (≥ 101 points) "Major" (worst injury). Injury severity quantified using MHISS is an important determinant of return to work after hand or forearm injury
Standard Hydraulic JAMAR dynamometer (Bellace, Healy, Besser, Byron, & Hohman, 2000), and Pinch Gauge (Radomski & Latham, 2008). A change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2).
  It Measures grip and pinch strength ,respectively.
Semmes-Weinstein Monofilament Test(van Vliet, Novak, & Mackinnon, 1993). a change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2).
  Measures low threshold of touch perception on an ordinal scale
Visual Analog Scale. A change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  Pain
Return -to-work self-efficacy scale-19 (RTWSE-19). (Shaw, Reme, Linton, Huang, & Pransky, 2011). Arabic version | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  The 19-item return-to-work self-efficacy (RTWSE-19) scale is a self-report measure intended to assess workers' beliefs of their current ability to resume normal job responsibilities following pain onset. Scores range from 1-10 which is obtained by summing all item scores and divide them by 19.
The Employment Barriers Questionnaire (EBQ) (Ratzon, Starik, Huber, & Zeilig, 2019). A change is being assessed. | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  A self-report questionnaire that aims to identify: 1. Potential work environment and job tasks obstacles 2. Overall level of restriction drawn by the obstacles, 3. Subjects' perception of the possibilities to make adaptations (PPMA) that might make work more accessible. The questionnaire is composed of 67 items separated into two parts. The first part assesses possible environmental barriers. The second part assesses possible job task barriers (including task limitations) in three categories: physical, cognitive and communication barriers. In each category, the items are measured by level of restriction scale (0 to 4) and PPMA (yes/no/no need for adaptation). In the second part, the frequency of the task is also estimated (0 to 4). Finally, two items assess the perception of the person on the extent of the employer's cooperation and the need for therapeutic mediation.
The Readiness for Return-to-Work (RRTW) scale (Franche, Corbière, Lee, Breslin, & Hepburn, 2007). A change is being assessed | Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  The Readiness for RTW scale is developed and validated in a Canadian cohort study it consist of 13 questions for people not working which includes Precontemplation, Contemplation, prepared for action (self-evaluative and behavioral) and 9 questions for people working which include Uncertain maintenance and Proactive maintenance. Psychometric properties of the newly developed instrument suggest that the application of the Readiness for Change model to return-to-work is relevant to work disability research. Confirmatory factor analyses had satisfactory fit indices to confirm the initial model.
Return-to-work status questionnaire (Boyle, Cassidy, & Côté, 2019). A change is being assessed | Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  A self-report return to work measure RTW at baseline and follow up. The baseline questionnaire has 24-items and elicits the following information: date of injury, days off because of the injury, current work status, reasons for not working and claim-related questions. The follow-up questionnaire is composed of 12- items addressing current working status, expectations for returning to work and reasons for not working. Nine of the items in the follow-up questionnaire are the same as the baseline questionnaire and five of them are used to generate the return-to-work status.The participant's return-to-work status could be defined as working with no modifications, working with modifications, tried to go back to work, in labor market retraining (LMR), gone back to school, or not working
Work Behavior inventory (G. Bryson, M. D. Bell, P. Lysaker, & W. J. P. R. J. Zito, 1997b). A change is being assessed | Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  The Work Behavior Inventory (WBI) is a standardized work performance assessment instrument specifically designed for people with severe mental illness. Test construction employed rational and empirical approaches yielding a 36-item inventory with five scales. It assesses vocational functioning for people with severe mental illness. It is rated in a work setting by an employment specialist through observation and an interview with the immediate supervisor.(Bull et al., 2015).
Post Traumatic Growth Inventory (PTGI) (Tedeschi & Calhoun, 1996). A change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  An instrument for assessing positive outcomes reported by persons who have experienced traumatic events. This 21-item scale includes factors of New Possibilities, Relating to Others, Personal Strength, Spiritual Change, and Appreciation of Life
The 12-item WHODAS 2.0 questionnaire - Arabic(Badr and Abd El Aziz 2007; Üstün et al. 2010). A change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  Measurement of health status. Provides a summering measure of functioning and disability that is reliable and valid across geographic regions, diagnostic groups, ages and genders. Can measure severity, monitor impact of programs, determine the score of individuals or groups in relation to the general population, or compare groups with respect to their disability. Explores what people do in different areas of life. All domains are mapped directly on ICF's activity and participation component: cognition, mobility, self-care, interpersonal interaction, life activities, and participation in society.
The Medical Outcome Study Short Form 12 (Ware Jr, Kosinski, & Keller, 1996). A change is being assessed | Baseline Time (T1), Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  This short version of the SF-36 tool consists of 12 items and eight scales: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and perceived mental health (MH). It has 35 possible response choice indicator variables; for example, the physical functioning item has three response choice categories, 1(yes, limited a lot), 2 (yes, limited a little), 3 (no, not limited at all). The composite physical (PCS) and mental health (MCS) scores are computed using the scores of the 12 items, ranging from 0 to 100, where zero reflects the lowest health level and 100 the highest level
Single Subject Job Satisfaction Scale (Dolbier et al. 2005). A change is being assessed | Discharge 4-6 weeks (T2), 3 months (T3), 6 months (T4) , 9 months (T5).
  single-item assessment tool, that is, whether or not the participant was satisfied with his/her a) current job and b) family life. Satisfaction items were scored on a four-point Likert scale with an option of 1) satisfied, 2) fairly satisfied, 3) fairly dissatisfied, and 4) dissatisfied. It was reversely scored so that higher score indicates a higher level of satisfaction. These items were taken from the Brief Job Stress Questionnaire, The items have been frequently used in past studies to measure job and family satisfaction at the workplaces14-16). The test-retest stability over 1 yr with job and life satisfaction was rs=0.468 and rs=0.567, respectively (p<0.001).

CONTACTS AND LOCATIONS:
Overall Officials: Navah Z Ratzon, Professor, Principal Investigator — Tel Aviv University
Locations (1):
- Arab American University, Jenin, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No